CLINICAL TRIAL: NCT02380820
Title: Comparative Measurements of Interface Pressures Between Two Pressure-ulcer Prevention Mattresses: Softform Premier and Airsoft Duo
Acronym: SPA2-INVACARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Invacare Poirier S.A.S. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2014/CEDMH-01; 2014-A01214-43 (Other: RCB number)
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Pressure Ulcer
Keywords: Mattress; Preventing bed sores; Skin pressure
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AirsoftDuo first (Experimental): Patients randomized to this arm will be placed on the Airsoft Duo mattress, and the investigator will proceed with 2 series (for reproductibility) of measures for 30 minutes with the bed headboard at 0°. A pause, consisting of ten minutes of sitting and 1 minute of verticalization is then carried out. The bed is then positioned at 30°, and the 2 series of measures over 30 minutes are repeated. The next day, all of the above are repeated with the Softform Premium mattress (in static mode). The patient will then continue his/her stay with the Softform Premium mattress (in static mode) for 1 month.
  Intervention: Airsoft Duo mattress Intervention: Softform Premier mattress (in static mode)
  Interventions: Device: Airsoft Duo mattress; Device: Softform Premier mattress (in static mode)
- Softform Premium first (Experimental): Patients randomized to this arm will be placed on the Softform Premium mattress (in static mode), and the investigator will proceed with 2 series (for reproductibility) of measures for 30 minutes with the bed headboard at 0°. A pause, consisting of ten minutes of sitting and 1 minute of verticalization is then carried out. The bed is then positioned at 30°, and the 2 series of measures over 30 minutes are repeated. The next day, all of the above are repeated with the Airsoft Duo mattress. The patient will then continue his/her stay with the Airsoft Duo mattress for 1 month.
  Intervention: Softform Premier mattress (in static mode) Intervention: Airsoft Duo mattress
  Interventions: Device: Airsoft Duo mattress; Device: Softform Premier mattress (in static mode)

INTERVENTIONS:
Device: Airsoft Duo mattress — A multi-layer mattress for pressure sore prevention. Made by NAUER FOAMPARTNER AG et OBA AG (Germany).
Device: Softform Premier mattress (in static mode) — A multi-layer mattress for pressure sore prevention. Made by INVACARE MSS (United Kingdom).

SUMMARY:
The main objective of this study is to compare the Softform Premier mattress (in static mode) and AIRSOFT DUO mattresses in terms of skin pressures measured at the sacral area.

DETAILED DESCRIPTION:
The secondary objectives of the study are to compare the two devices in terms of:

A. contact surface. B. heel pressure. C. On the occurrence of pressure ulcers anywhere on the body at month 1. D. patient comfort after 1 month (visual analog scale ranging from 1 to 10).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient spends more than 12 hours in bed with a possible verticalization and a predictable length of stay of at least 1 month.
* The patient has a stable medical condition (no complications in the last 10 days) without pressure ulcers
* The patient is at risk of pressure ulcers assessed a score ≤ 14 on the Norton scale
* The patient's weight is less than 120 Kg

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Contra-indication for strict decubitus dorsal position
* The patient has a rotation of the pelvis, asymmetric deformations of the hips in the frontal plane.
* The patient has bedsores, a recent scar in a pressure area.
* The patient has a knee flexion deformity> 10 °
* The patient is agitated or uncooperative
* The patient's weight is greater than 120 Kg

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Interface pressure in the sacral zone (mm Hg) as measured by a Model X3 sensor pressure captor sheet | Day 1

SECONDARY OUTCOMES:
Contact surface area (cm^2) as measured by a Model X3 sensor pressure captor sheet | Day 1
Interface pressure at the heel (mm Hg) as measured by a Model X3 sensor pressure captor sheet | Day 1
Presence/absence of a pressure ulcer over the past month | 1 month
Patient-rated comfort as measured by the visual analog scale | 1 month
  Visual analog scale ranging from 0 to 10

OTHER OUTCOMES:
Age (years) | Baseline (Day 0)
Sex (F/M) | Baseline (Day 0)
Weight (kg) | Baseline (Day 0)
Height (cm) | Baseline (Day 0)
Body mass index (kg/m^2) | Baseline (Day 0)
Norton risk score | Baseline (Day 0)
Albuminemia | Baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Viollet, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - EHPAD La Chimotaie, Cugan Montaigu Cedex
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - EHPAD Notre Dame des Pins, Saint-Privat-des-Vieux